CLINICAL TRIAL: NCT02498457
Title: The First Affiliated Hospital of Chongqing Medical University
Brief Title: The Effects and Safety of Low Calcium Dialysis on Coronary Artery Calcification in Maintenance Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yunfeng Xia, Department of Nephrology, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1stChongqingMU snkxia1
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Coronary Artery Calcification
Keywords: maintenance hemodialysis patients; coronary artery calcification; low calcium dialysate; effects; safety

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low calcium dialysis (Active Comparator): patients in this group will be dialyzed using a dialysate with a calcium concentration 1.25mmol/L.
  Interventions: Other: low calcium dialysis
- Routine dialysis (Other): Patients in this groups will be dialyzed using routine dialysate with a calcium concentration 1.5mmol/L.
  Interventions: Other: low calcium dialysis

INTERVENTIONS:
Other: low calcium dialysis — patients in this group will receive low calcium dialysis for 1 year.

SUMMARY:
This study aim to observe the preventive effect and the long term safety of low calcium dialysis on coronary artery calcification in Maintenance hemodialysis (MHD) patients.

DETAILED DESCRIPTION:
MHD patients recruited in this study were randomly divided into two groups: routine dialysis group (with dialysate calcium concentration 1.5mmol/L) and low calcium dialysis group (with dialysate calcium concentration 1.25mmol/L). All patients were dialyzed thrice weekly for 4 hours with a bicarbonate-based solution. They were followed up in every dialysis interview during the 1-year study, the occurrence of all adverse reactions associated with dialysis were recorded during the study. All patients received heart spiral CT examination before and at the end of the study. Coronary artery calcification was assessed by a certain professional who was not affiliated to the dialysis center.

ELIGIBILITY:
Inclusion Criteria:

* Maintenance hemodialysis (MHD) patients who dialyze thrice weekly in our hospital with serum iPTH <500pg/ml, adjusted serum calcium≧8.4mg/dl in two serial tests.
* Patients who have no chronic infection or malignant tumour and with relatively stable heart and lung function.
* Patients who signed informed consent documents at the time of enrollment in the study.

Exclusion Criteria:

* Patients whose heart or lung function are poor, or with unstable hemodynamics.
* Patients who are diagnosed active pulmonary tuberculosis, AIDS, malignant tumour, or decompensated liver cirrhosis.
* Patients who are unable or unwilling to cooperate with the researchers in the treatment and follow-up.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Changes in coronary artery calcification after 1 year's treatment | 1 year

SECONDARY OUTCOMES:
The intolerance of low calcium dialysis because of adverse reactions associated with dialysis were recorded during the study | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hua Gan, Dr., Study Director — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China